CLINICAL TRIAL: NCT03831308
Title: Evaluating, Following, and Supporting Breast Cancer Patients in a Better Way
Brief Title: Evaluating and Following Breast Cancer Patients in a Better Way
Acronym: EFBCancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centro Hospitalar Lisboa Ocidental (Other Government)
Collaborators: University of Lisbon (Other)
Responsible Party: Principal Investigator, Vasco Fonseca, Dr, Centro Hospitalar Lisboa Ocidental
Other Study IDs: CentroHLO_EFBreastCancer
Record Dates: First submitted 2018-11-15; First posted 2019-02-05 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Breast Cancer Female
Keywords: Breast cancer; Physical exercise and Breast Cancer; Cognitive status and Breast Cancer; Physical activity and quality of life of cancer patients; New tools for evaluating breast Cancer patients
MeSH Terms: conditions — Breast Neoplasms; Motor Activity | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breast cancer new diagnosis: group will include volunteer women, diagnosed with breast cancer, in any stage, aged 18y or more; at least 100 patients will be recruited in medical oncology appointments; all subjects should be periodically submitted to non-invasive evaluation tests - that is, clinical test/clinical and physical assessment to collect information on fitness status, lifestyle, cognitive and psychological status, bone's health and quality of life
  Interventions: Diagnostic Test: clinical and physical assessment

INTERVENTIONS:
Diagnostic Test: clinical and physical assessment — information will be collected on fitness status, lifestyle, cognitive and psychological status, bone's health and quality of life

SUMMARY:
The current observational study aims at analysing current semiology on breast cancer patients aiming at noting indicators and signs with significant relationship with the disease outcomes.

To reach the primary objective, of identifying most prominent indicators and signs, a study group of at least 100 female patients with breast cancer diagnosis will be recruited to participate voluntarily. The study group will include at least 20 patients with metastatic cancer and 30 patients with indication to adjuvant chemotherapy. Their physical activity habits and lifestyle will be noted. The observational study will consist in the periodic registration of the overall physical and psychological condition. The variables and tests below will be measured and registered, periodically:

* periodical assessment of the quality of life
* periodical assessment of the fitness status of the subjects
* assessment of changes in bone density/progression of osteoporosis
* assessment of changes in cognitive function
* assessment of sleep disorders

The collected results will be statistically analysed, in order to:

* Identify variables that are statistically significantly different from expected values
* quantify statistically significant differences, whenever possible

The results will be used to better describe the breast cancer population

DETAILED DESCRIPTION:
Breast Cancer treatment is expected to have the best outcome when adapted to the patients' health, and physical condition. The investigators aim at contributing to produce an improved algorithm to evaluate breast cancer patients.

The semiologic evaluation of patients is changing, as a result of scientific advances, easier and rapid access to information, the incorporation of ICT (information and communication technologies) etc. Profound changes are expected, namely in incorporating new technologies to improve patient's evaluation.

Medicine is also called to give better support to cancer patients, which disease is not active but may evolve in the future. Cancer is more and more regarded as a chronic ailment, as the acute life-threatening conditions are fortunately becoming less and less frequent. In these cases, medicine is requested to provide ways of improving longevity with quality of life. Physical activity may play an important role in achieving such a goal. The investigators think that possibly the same kind of approach, i.e. considering physical activity, although to a different extent, should also be considered in the case of some patients with active disease. Human relationships play a very important role in supporting the patients' wellness, in impacting their quality of life, and in ensuring that the patients have the most adequate treatment, taking into account their true health conditions.

This change of paradigm in Medicine is very important in areas as Oncology. Clinicians need new tools to give the best treatment to patients. These new tools will certainly soon incorporate new technologies that will call for different patterns of patients' validation.

The question to be answered is if whether or not the introduction of new variables for the assessment of disease progression/quality of life of breast cancer patients and survivors will help improve medical reasoning of the general condition of the patient.

As future goals, subsequently to the present observational study, the investigators look forward to provide answers to:

* what kind of physical and cognitive evaluation should be offered to Breast Cancer Patients?
* How can existing knowledge on physical motility be incorporated in the clinical practice? Namely in physical, and cognitive evaluation? (and finally assessing if such evaluation has practical impact) Moreover, the extended data set, expected to be obtained in the current study, is likely to be useful in developing strategies to motivate patients to follow an active lifestyle and balanced diet, as well as in helping adapt interventions that aim at improving survival rates and the quality of life.

The relevant observations, summarized in this study, are expected to positively act on semiology evaluation of the breast cancer patients on daily medical practice, through an improved algorithm. Such algorithm should be suitable for the clinical practice and compatible with artificial intelligence tools.

ELIGIBILITY:
Inclusion Criteria:

* women
* age > 18y
* diagnosed with breast cancer

Exclusion Criteria:

* men
* informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Although it may occur, breast cancer is rare in men
Study Population: women with breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Global medical assessment | 1st month at enrolment
  during the first medical appointment general health status and cancer staging will be noted for each participant; participants will be asked about their lifestyle, namely to register those with a sedentary lifestyle vs those enrolled in any regular physical activity
Assessment of changes in the cardiac function/fitness status of the subjects | 1st month at enrolment, 6 and 12 months after enrolment
  The modified Bruce Protocol is a cardiac stress test that includes 2 warmup stages, each lasting 3 minutes and aims at evaluate the cardiac function will be collected, assessed and registered according to current clinical practice

SECONDARY OUTCOMES:
screening sleep disorders and assessing changes in sleeping patterns | 1st month at enrolment, 6 and 12 months after enrolment
  A validated questionnaire to assist the screening of sleep disorders will be periodically applied; such questionnaire consists in 16 questions graded from 1=never to 5=always, with an interpretation guide to track the diagnostic domains: insomnia, psychiatric disorders, circadian rhythm disorder, movement disorders, and parasomnias
Assessment of changes in bone's density | 1st month at enrolment, 6 and 12 months after enrolment
  Bone Densitometry - Bone densitometry (or DEXA) uses a very small dose of radiation to measure bone density and bone loss. The test can help determine any advancement of osteoporosis.
Assessment of changes in the cognitive function | 1st month at enrolment, 6 and 12 months after enrolment
  Mini-Mental State Examination (MMSE) or Folstein test is a 30-point questionnaire that allows the examination of such functions as registration (repeating named prompts), attention and calculation, recall, language, ability to follow simple commands and orientation

CONTACTS AND LOCATIONS:
Overall Officials: Vasco Fonseca, Principal Investigator — Hospital S Francisco Xavier - Ocidental Lisbon Hospital Center, Lisbon, Portugal; Pedro Sarmento, PhD, Study Chair — Faculty of Human Motricity - University of Lisbon

IPD SHARING:
Plan to Share IPD: Undecided
undecided